CLINICAL TRIAL: NCT01925612
Title: A Phase 2 Study of Brentuximab Vedotin in Combination With Standard of Care Treatment (Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone [RCHOP]) or RCHP (Rituximab, Cyclophosphamide, Doxorubicin, and Prednisone) as Front-line Therapy in Patients With Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: Study of Brentuximab Vedotin Combined With RCHOP or RCHP in Front-line Treatment of Patients With Diffuse Large B-cell Lymphoma (DLBCL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision based on portfolio prioritization and changing treatment landscape in frontline DLBCL
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGN35-017
Record Dates: First submitted 2013-08-15; First posted 2013-08-20 (Estimated); Results first posted 2018-06-21 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-05

CONDITIONS: Lymphoma, B-cell; Lymphoma, Large B-cell, Diffuse
Keywords: Antibodies, Monoclonal; Antibody-Drug Conjugate; Antigens, CD30; Drug Therapy; Hematologic Diseases; Lymphoma, B-cell; Lymphoma, Large B-cell, Diffuse; Monomethyl auristatin E
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Hematologic Diseases | interventions — Brentuximab Vedotin; Rituximab; Vincristine; Cyclophosphamide; Prednisone; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part 1: BV(1.2 mg/kg) + RCHOP (Experimental): Brentuximab vedotin 1.2 mg/kg plus rituximab, cyclophosphamide, doxorubicin, vincristine, prednisone
  Part 1 of the study is a phase 2, randomized, open-label, multicenter study designed to evaluate the antitumor activity and safety of brentuximab vedotin when administered in combination with standard RCHOP chemotherapy (rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone). Patients in this arm were randomized into the 1.2 mg/kg brentuximab vedotin dosing cohort, to be administered in combination with RCHOP.
  Interventions: Drug: brentuximab vedotin; Drug: rituximab; Drug: vincristine; Drug: cyclophosphamide; Drug: prednisone; Drug: doxorubicin
- Part 1: BV(1.8 mg/kg) + RCHOP (Experimental): Brentuximab vedotin 1.8 mg/kg plus rituximab, cyclophosphamide, doxorubicin, vincristine, prednisone
  Part 1 of the study is a phase 2, randomized, open-label, multicenter study designed to evaluate the antitumor activity and safety of brentuximab vedotin when administered in combination with standard RCHOP chemotherapy (rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone). Patients in this arm were randomized into the 1.8 mg/kg brentuximab vedotin dosing cohort, to be administered in combination with RCHOP.
  Interventions: Drug: brentuximab vedotin; Drug: rituximab; Drug: vincristine; Drug: cyclophosphamide; Drug: prednisone; Drug: doxorubicin
- Part 2: BV(1.8 mg/kg) + RCHP (Experimental): Brentuximab vedotin 1.8 mg/kg plus rituximab, cyclophosphamide, doxorubicin, prednisone
  Part 2 of the study is a phase 2, non-randomized, open-label, multicenter study designed to evaluate the antitumor activity and safety of brentuximab vedotin 1.8 mg/kg when administered in combination with RCHP chemotherapy (rituximab, cyclophosphamide, doxorubicin, and prednisone). Patients in this treatment arm were enrolled into a dosing cohort with 1.8 mg/kg brentuximab vedotin administered in combination with RCHP.
  Interventions: Drug: brentuximab vedotin; Drug: rituximab; Drug: cyclophosphamide; Drug: prednisone; Drug: doxorubicin
- Part 3: RCHOP (Active Comparator): Rituximab, cyclophosphamide, doxorubicin, vincristine, prednisone
  Part 3 of the study is a phase 2, randomized, open-label, multicenter study designed to evaluate the antitumor activity and safety of brentuximab vedotin 1.8 mg/kg when administered in combination with RCHP chemotherapy compared to RCHOP chemotherapy alone. Patients in this treatment arm were randomized to receive RCHOP treatment alone.
  Interventions: Drug: rituximab; Drug: vincristine; Drug: cyclophosphamide; Drug: prednisone; Drug: doxorubicin
- Part 3: BV(1.8 mg/kg) + RCHP (Experimental): Brentuximab vedotin 1.8 mg/kg plus rituximab, cyclophosphamide, doxorubicin, prednisone
  Part 3 of the study is a phase 2, randomized, open-label, multicenter study designed to evaluate the antitumor activity and safety of brentuximab vedotin 1.8 mg/kg when administered in combination with RCHP chemotherapy compared to RCHOP chemotherapy alone. Patients in this treatment arm were randomized to receive RCHOP treatment alone. Randomization in this part of the study is for the purpose of evaluating the safety of 1.8 mg/kg brentuximab vedotin in combination with RCHP versus standard RCHOP chemotherapy.
  Part 3 of the study is a phase 2, randomized, open-label, multicenter study designed to evaluate the antitumor activity and safety of brentuximab vedotin 1.8 mg/kg when administered in combination with RCHP chemotherapy compared to RCHOP chemotherapy alone. Patients in this treatment arm were randomized to receive 1.8 mg/kg brentuximab vedotin administered in combination with RCHP.
  Interventions: Drug: brentuximab vedotin; Drug: rituximab; Drug: cyclophosphamide; Drug: prednisone; Drug: doxorubicin

INTERVENTIONS:
Drug: brentuximab vedotin — 1.2 mg/kg by IV infusion every 3 weeks for up to 6 cycles
  Other Names: Adcetris, SGN-35
  Arms: Part 1: BV(1.2 mg/kg) + RCHOP
Drug: brentuximab vedotin — 1.8 mg/kg by IV infusion every 3 weeks for up to 6 cycles
  Other Names: Adcetris, SGN-35
  Arms: Part 1: BV(1.8 mg/kg) + RCHOP; Part 2: BV(1.8 mg/kg) + RCHP; Part 3: BV(1.8 mg/kg) + RCHP
Drug: rituximab — 375 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
Drug: vincristine — 1.4 mg/m2 every 3 weeks by IV infusion for up to 6 cycles (dose capped at 2 mg total)
  Arms: Part 1: BV(1.2 mg/kg) + RCHOP; Part 1: BV(1.8 mg/kg) + RCHOP; Part 3: RCHOP
Drug: cyclophosphamide — 750 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
Drug: prednisone — 100 mg on Days 1 to 5 of each 3-week cycle, orally for up to 6 cycles
Drug: doxorubicin — 50 mg/m2 every 3 weeks by IV infusion for up to 6 cycles

SUMMARY:
This study has 3 parts. The purpose of Part 1 of this study is to assess the safety and efficacy of brentuximab vedotin in combination with RCHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone) (known as BV+RCHOP) in patients with DLBCL who have never been treated. Patients will be randomly assigned in a 1:1 ratio to receive RCHOP together with 1 of 2 doses of brentuximab vedotin. Patients will be tested to see if there is a difference in side effects between the 2 groups.

The purpose of Part 2 of this study is to assess the safety and efficacy of brentuximab vedotin in combination with RCHP (rituximab, cyclophosphamide, doxorubicin, and prednisone) (known as BV+RCHP) in patients with CD30-positive DLBCL who have never been treated. Patients will be enrolled to receive RCHP together with 1.8mg/kg of brentuximab vedotin.

The purpose of Part 3 of this study is to assess the safety and efficacy of BV+RCHP compared to standard RCHOP in patients with CD30-positive DLBCL that have never been treated. Patients will be randomly assigned in a 1:1 ratio to receive either BV+RCHP or RCHOP. Patients will be tested to see if there is a difference in side effects between the 2 groups.

DETAILED DESCRIPTION:
In the first part of this study, patients in the 2 groups were tested to see if there was a difference in the response to treatment and whether there were differences in the side effects (unwanted effects).

The second and third parts of the study are being done to see if there are any side effects (unwanted effects) of the higher dose of brentuximab vedotin when combined with a modified version of RCHOP that omits vincristine. The third part of the study is being done to see if there is a difference between BV+RCHP and RCHOP in the response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naive patients with systemic de novo or transformed diffuse large B cell lymphoma (DLBCL) or follicular non-Hodgkin lymphoma (NHL) grade 3b
* International Prognostic Index (IPI) score greater than or equal to 3 for patients greater than 60 years of age or age-adjusted IPI (aaIPI) score of 2 or 3 for patients less than or equal to 60 years of age
* Stage IAX (bulk defined as single lymph node mass >10 cm in diameter), IB-IV disease
* Measurable disease of at least 1.5 cm
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Patients in Parts 2 and 3 must have histologically confirmed diagnosis of CD30-positive DLBCL

Exclusion Criteria:

* Previous history of treated indolent lymphoma
* History of another primary malignancy that has not been in remission for 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2013-08; Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Ruffner, Study Director — Seagen Inc.
Locations (51):
- United States (36):
  - Arizona Oncology Associates, PC - HAL, Phoenix, Arizona
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - City of Hope National Medical Center, Duarte, California
  - Sansum Clinic, Santa Barbara, California
  - Stanford Cancer Center, Stanford, California
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - Augusta University, Augusta, Georgia
  - Cardinal Bernardin Cancer Center / Loyola University Medical Center, Maywood, Illinois
  - Illinois Cancer Specialists / Advocate Lutheran General Hospital, Niles, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic Cancer Research, Billings, Montana
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Summit Medical Group, Morristown, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - New York Oncology Hematology, P.C., Albany, New York
  - Mid Ohio Oncology/Hematology Inc, Columbus, Ohio
  - Willamette Valley Cancer Institute and Research Center, Springfield, Oregon
  - Northwest Cancer Specialists, P.C., Tualatin, Oregon
  - Saint Francis Hospital / Bon Secours, Greenville, South Carolina
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Texas Oncology - Austin Midtown, Austin, Texas
  - Texas Oncology - Baylor Sammons Cancer Center, Dallas, Texas
  - US Oncology Investigational Products Center (IPC), Fort Worth, Texas
  - MD Anderson Cancer Center / University of Texas, Houston, Texas
  - Texas Oncology - San Antonio Medical Center, San Antonio, Texas
  - US Oncology Central Regulatory, The Woodlands, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Benaroya Research Institute/Virginia Mason Medical Center, Seattle, Washington
- Czechia (4):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove-oddeleni klinicke hematologie, Hradec Králové
  - Fakultni Nemocnice Kralovske Vinohrady, Prague
  - Fakultni nemocnice v Motole, Prague
- Italy (4):
  - Centro di Riferimento Oncologico di Aviano, Aviano
  - Instituto di Ematologia ed Oncologia Medica, Bologna
  - Azienda Ospedaliero-Universitaria Pisana - Ospedale S. Chiara, Pisa
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
- Poland (3):
  - COPERNICUS Podmiot Leczniczy Sp. z o.o. Wojewodzkie Centrum Onkologii, Gdansk
  - Malopolskie Centrum Medyczne S.C., Krakow
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Ministerstwa Spraw Wewnetrznych z Warminsko-Mazurskim, Olsztyn
- Spain (4):
  - Hospital de la Santa Creu i Sant Paul, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Institut Català D'oncologia, L'Hospitalet de Llobregat
  - Complejo Hospitalano de Navarra Servicio Hematologia, Pamplona

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two patients enrolled but did not receive treatment.
Groups:
- Part 1: BV(1.2 mg/kg) + RCHOP: Part 1 of the study is randomized and open-label. Brentuximab vedotin was administered at 1.2mg/kg in combination with standard RCHOP chemotherapy (rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone).
  brentuximab vedotin: 1.2 mg/kg by IV infusion every 3 weeks for up to 6 cycles
  rituximab: 375 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
  vincristine: 1.4 mg/m2 every 3 weeks by IV infusion for up to 6 cycles (dose capped at 2 mg total)
  cyclophosphamide: 750 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
  prednisone: 100 mg on Days 1 to 5 of each 3-week cycle, orally for up to 6 cycles
  doxorubicin: 50 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
- Part 1: BV(1.8 mg/kg) + RCHOP: Part 1 of the study is a randomized and open-label. Brentuximab vedotin was administered at 1.8 mg/kg in combination with standard RCHOP chemotherapy (rituximab, cyclophosphamide, doxorubicin, vincristine, and prednisone).
  brentuximab vedotin: 1.8 mg/kg by IV infusion every 3 weeks for up to 6 cycles
  rituximab: 375 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
  vincristine: 1.4 mg/m2 every 3 weeks by IV infusion for up to 6 cycles (dose capped at 2 mg total)
  cyclophosphamide: 750 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
  prednisone: 100 mg on Days 1 to 5 of each 3-week cycle, orally for up to 6 cycles
  doxorubicin: 50 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
- Part 2: BV(1.8 mg/kg) + RCHP: Part 2 of the study was non-randomized and open-label. Brentuximab vedotin (1.8 mg/kg) was administered in combination with RCHP chemotherapy (rituximab, cyclophosphamide, doxorubicin, and prednisone).
  brentuximab vedotin: 1.8 mg/kg by IV infusion every 3 weeks for up to 6 cycles
  rituximab: 375 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
  cyclophosphamide: 750 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
  prednisone: 100 mg on Days 1 to 5 of each 3-week cycle, orally for up to 6 cycles
  doxorubicin: 50 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
- Part 3: BV(1.8 mg/kg) + RCHP: Part 3 of the study was randomized and open-label. Brentuximab vedotin (1.8 mg/kg) was administered in combination with RCHP chemotherapy.
  brentuximab vedotin: 1.8 mg/kg by IV infusion every 3 weeks for up to 6 cycles
  rituximab: 375 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
  cyclophosphamide: 750 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
  prednisone: 100 mg on Days 1 to 5 of each 3-week cycle, orally for up to 6 cycles
  doxorubicin: 50 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
- Part 3: RCHOP: Part 3 of the study was randomized and open-label. RCHOP chemotherapy was administered alone.
  rituximab: 375 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
  vincristine: 1.4 mg/m2 every 3 weeks by IV infusion for up to 6 cycles (dose capped at 2 mg total)
  cyclophosphamide: 750 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
  prednisone: 100 mg on Days 1 to 5 of each 3-week cycle, orally for up to 6 cycles
  doxorubicin: 50 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
Period: Overall Study
Arm/Group | Part 1: BV(1.2 mg/kg) + RCHOP | Part 1: BV(1.8 mg/kg) + RCHOP | Part 2: BV(1.8 mg/kg) + RCHP | Part 3: BV(1.8 mg/kg) + RCHP | Part 3: RCHOP
Started | 29 | 22 | 11 | 11 | 12
Completed | 25 | 18 | 10 | 10 | 10
Not Completed | 4 | 4 | 1 | 1 | 2
Not completed — Progressive Disease | 1 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 3 | 3 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Part 1: BV(1.2 mg/kg) + RCHOP: Brentuximab vedotin 1.2 mg/kg plus rituximab, cyclophosphamide, doxorubicin, vincristine, prednisone
  brentuximab vedotin: 1.2 mg/kg by IV infusion every 3 weeks for up to 6 cycles
  rituximab: 375 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
  vincristine: 1.4 mg/m2 every 3 weeks by IV infusion for up to 6 cycles (dose capped at 2 mg total)
  cyclophosphamide: 750 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
  prednisone: 100 mg on Days 1 to 5 of each 3-week cycle, orally for up to 6 cycles
  doxorubicin: 50 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
- Part 1: BV(1.8 mg/kg) + RCHOP: Brentuximab vedotin 1.8 mg/kg plus rituximab, cyclophosphamide, doxorubicin, vincristine, prednisone
  brentuximab vedotin: 1.8 mg/kg by IV infusion every 3 weeks for up to 6 cycles
  rituximab: 375 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
  vincristine: 1.4 mg/m2 every 3 weeks by IV infusion for up to 6 cycles (dose capped at 2 mg total)
  cyclophosphamide: 750 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
  prednisone: 100 mg on Days 1 to 5 of each 3-week cycle, orally for up to 6 cycles
  doxorubicin: 50 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
- Part 2: BV(1.8 mg/kg) + RCHP; Part 3: BV(1.8 mg/kg) + RCHP: Brentuximab vedotin 1.8 mg/kg plus rituximab, cyclophosphamide, doxorubicin, prednisone
  brentuximab vedotin: 1.8 mg/kg by IV infusion every 3 weeks for up to 6 cycles
  rituximab: 375 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
  cyclophosphamide: 750 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
  prednisone: 100 mg on Days 1 to 5 of each 3-week cycle, orally for up to 6 cycles
  doxorubicin: 50 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
- Part 3: RCHOP: Rituximab, cyclophosphamide, doxorubicin, vincristine, prednisone
  rituximab: 375 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
  vincristine: 1.4 mg/m2 every 3 weeks by IV infusion for up to 6 cycles (dose capped at 2 mg total)
  cyclophosphamide: 750 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
  prednisone: 100 mg on Days 1 to 5 of each 3-week cycle, orally for up to 6 cycles
  doxorubicin: 50 mg/m2 every 3 weeks by IV infusion for up to 6 cycles
- Total: Total of all reporting groups
Arm/Group | Part 1: BV(1.2 mg/kg) + RCHOP | Part 1: BV(1.8 mg/kg) + RCHOP | Part 2: BV(1.8 mg/kg) + RCHP | Part 3: BV(1.8 mg/kg) + RCHP | Part 3: RCHOP | Total
Number analyzed (Participants) | 29 | 22 | 11 | 11 | 12 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 7 | 5 | 6 | 39
  >=65 years | 19 | 11 | 4 | 6 | 6 | 46
Age, Continuous [Median (Full Range); unit: years] | 70 [33 to 80] | 64 [21 to 81] | 59 [22 to 78] | 68 [46 to 74] | 65 [41 to 80] | 66 [21 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 4 | 10 | 6 | 39
  Male | 16 | 16 | 7 | 1 | 6 | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 1 | 0 | 1 | 8
  Not Hispanic or Latino | 25 | 18 | 8 | 11 | 11 | 73
  Unknown or Not Reported | 0 | 2 | 2 | 0 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 1 | 0 | 4
  White | 27 | 17 | 8 | 10 | 12 | 74
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 3 | 1 | 0 | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 29 | 22 | 11 | 8 | 10 | 82
  Czechia | 0 | 0 | 0 | 1 | 1 | 2
  Poland | 0 | 0 | 0 | 2 | 0 | 2
  Italy | 0 | 0 | 0 | 0 | 1 | 1
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — 0=Normal activity; 1=Symptoms but ambulatory; 2=In bed <50% of the time; 3= In bed >50% of the time; 4=100% bedridden; 5=Dead
  Participants
    0 | 5 | 4 | 1 | 4 | 4 | 18
    1 | 16 | 12 | 4 | 4 | 3 | 39
    2 | 8 | 6 | 6 | 3 | 5 | 28

OUTCOME MEASURES:

1. Primary Outcome: Complete Remission Rate
Description: Number (count) of participants that achieved remission according to the Revised Response Criteria for Malignant Lymphoma (Cheson 2007).
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: BV(1.2 mg/kg) + RCHOP | Part 1: BV(1.8 mg/kg) + RCHOP | Part 2: BV(1.8 mg/kg) + RCHP | Part 3: BV(1.8 mg/kg) + RCHP | Part 3: RCHOP
Number analyzed (Participants) | 29 | 22 | 11 | 11 | 12
Participants | 20 | 16 | 9 | 6 | 8

2. Primary Outcome: Incidence of Adverse Events
Description: Number (count) of participants that experienced at least 1 adverse event.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: BV(1.2 mg/kg) + RCHOP | Part 1: BV(1.8 mg/kg) + RCHOP | Part 2: BV(1.8 mg/kg) + RCHP | Part 3: BV(1.8 mg/kg) + RCHP | Part 3: RCHOP
Number analyzed (Participants) | 29 | 22 | 11 | 11 | 12
Participants | 29 | 22 | 11 | 11 | 12

3. Primary Outcome: Incidence of Laboratory Abnormalities
Description: Number (count) of participants that experienced a Grade 3 or higher maximum post-baseline laboratory toxicity (hematology and chemistry). Grades are defined using National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE), v4.03. Grade 1 = mild, no intervention needed; Grade 2 = moderate, minimal intervention needed; Grade 3 = severe or medically significant, hospitalization is required; Grade 4 = life-threatening, urgent intervention needed; Grade 5 = death related to adverse event.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: BV(1.2 mg/kg) + RCHOP | Part 1: BV(1.8 mg/kg) + RCHOP | Part 2: BV(1.8 mg/kg) + RCHP | Part 3: BV(1.8 mg/kg) + RCHP | Part 3: RCHOP
Number analyzed (Participants) | 29 | 22 | 11 | 11 | 12
Participants
  Any Hematology Test | 10 | 16 | 4 | 6 | 4
  Lymphocytes (x10^3/uL) | 8 | 15 | 3 | 4 | 4
  Absolute Neutrophil Count (x10^3/uL) | 4 | 4 | 1 | 2 | 0
  Neutrophils (x10^3/uL) | 4 | 4 | 1 | 2 | 0
  Leukocytes (x10^3/uL) | 3 | 2 | 1 | 1 | 1
  Hemoglobin (x10^3/uL) | 0 | 1 | 0 | 1 | 0
  Platelets (x10^3/uL) | 1 | 1 | 0 | 0 | 0
  Any Chemistry Test | 4 | 7 | 2 | 1 | 3
  Glucose (mg/dL) | 3 | 5 | 0 | 0 | 1
  Potassium (mEq)/L | 0 | 2 | 1 | 1 | 2
  Calcium (mg/dL) | 1 | 1 | 0 | 0 | 0
  Sodium (mEq/L) | 0 | 2 | 0 | 0 | 0
  Alanine Aminotransferase (IU/L) | 0 | 0 | 1 | 0 | 0

4. Secondary Outcome: Objective Response Rate
Description: Number (count) of participants that achieved complete or partial remission at the end of treatment according to the Revised Response Criteria for Malignant Lymphoma (Cheson 2007)
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: BV(1.2 mg/kg) + RCHOP | Part 1: BV(1.8 mg/kg) + RCHOP | Part 2: BV(1.8 mg/kg) + RCHP | Part 3: BV(1.8 mg/kg) + RCHP | Part 3: RCHOP
Number analyzed (Participants) | 29 | 22 | 11 | 11 | 12
Participants | 23 | 19 | 10 | 10 | 9

5. Secondary Outcome: Progression-free Survival
Description: Median progression-free survival (in months) and observed minimum-maximum range.
Time Frame: Up to approximately 4 years
Measure: Median (Full Range); unit: Months
Arm/Group | Part 1: BV(1.2 mg/kg) + RCHOP | Part 1: BV(1.8 mg/kg) + RCHOP | Part 2: BV(1.8 mg/kg) + RCHP | Part 3: BV(1.8 mg/kg) + RCHP | Part 3: RCHOP
Number analyzed (Participants) | 29 | 22 | 11 | 11 | 12
Months | NA [0.62 to 40.21] — Insufficient number of participants with events to determine median (<50%) | NA [1.28 to 39.85] — Insufficient number of participants with events to determine median (<50%) | NA [3.35 to 24.34] — Insufficient number of participants with events to determine median (<50%) | NA [3.25 to 15.41] — Insufficient number of participants with events to determine median (<50%) | NA [1.25 to 16.43] — Insufficient number of participants with events to determine median (<50%)

6. Secondary Outcome: Overall Survival
Description: Median overall survival (in months) and observed minimum-maximum range.
Time Frame: Up to approximately 4 years
Measure: Median (Full Range); unit: Months
Arm/Group | Part 1: BV(1.2 mg/kg) + RCHOP | Part 1: BV(1.8 mg/kg) + RCHOP | Part 2: BV(1.8 mg/kg) + RCHP | Part 3: BV(1.8 mg/kg) + RCHP | Part 3: RCHOP
Number analyzed (Participants) | 29 | 22 | 11 | 11 | 12
Months | NA [0.62 to 42.79] — Insufficient number of participants with events to estimate median (<50%) | NA [1.28 to 44.29] — Insufficient number of participants with events to estimate median (<50%) | NA [16.56 to 25.76] — Insufficient number of participants with events to estimate median (<50%) | NA [3.25 to 16.85] — Insufficient number of participants with events to estimate median (<50%) | NA [1.25 to 19.22] — Insufficient number of participants with events to estimate median (<50%)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from study Day 1 (predose) though the EOT visit or 30 days after the last study treatment (Brentuximab vedotin or combination treatment), whichever was later. However, all protocol-related AEs were collected from the time of informed consent.
Arm/Group | Part 1: BV(1.2 mg/kg) + RCHOP | Part 1: BV(1.8 mg/kg) + RCHOP | Part 2: BV(1.8 mg/kg) + RCHP | Part 3: BV(1.8 mg/kg) + RCHP | Part 3: RCHOP
All-Cause Mortality (participants affected / at risk) | 1/29 | 2/22 | 0/11 | 1/11 | 2/12
Serious Adverse Events (participants affected / at risk) | 16/29 | 14/22 | 5/11 | 4/11 | 4/12
Other Adverse Events (participants affected / at risk) | 29/29 | 22/22 | 11/11 | 11/11 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: BV(1.2 mg/kg) + RCHOP (N=29) | Part 1: BV(1.8 mg/kg) + RCHOP (N=22) | Part 2: BV(1.8 mg/kg) + RCHP (N=11) | Part 3: BV(1.8 mg/kg) + RCHP (N=11) | Part 3: RCHOP (N=12)
Febrile Neutropenia (Blood and lymphatic system disorders) | 8 (13) | 8 (13) | 2 (2) | 0 (0) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pantoea agglomerans infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenic colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Guillain-barre syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stevens-johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: BV(1.2 mg/kg) + RCHOP (N=29) | Part 1: BV(1.8 mg/kg) + RCHOP (N=22) | Part 2: BV(1.8 mg/kg) + RCHP (N=11) | Part 3: BV(1.8 mg/kg) + RCHP (N=11) | Part 3: RCHOP (N=12)
Nausea (Gastrointestinal disorders) | 14 (24) | 15 (23) | 8 (9) | 4 (6) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 14 (19) | 15 (23) | 3 (4) | 6 (8) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (9) | 9 (12) | 6 (6) | 1 (1) | 5 (5)
Vomiting (Gastrointestinal disorders) | 7 (9) | 14 (17) | 2 (2) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 8 (10) | 3 (4) | 3 (3) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 4 (5) | 3 (3) | 1 (2) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tongue discolouration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (6) | 9 (10) | 8 (10) | 3 (3) | 3 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (2) | 2 (2) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (3) | 3 (3) | 1 (2) | 1 (1) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 17 (28) | 16 (30) | 7 (7) | 2 (2) | 3 (4)
Asthenia (General disorders) | 8 (19) | 7 (8) | 0 (0) | 0 (0) | 2 (3)
Chills (General disorders) | 7 (12) | 4 (4) | 3 (3) | 1 (2) | 0 (0)
Oedema peripheral (General disorders) | 7 (9) | 7 (8) | 1 (2) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 6 (9) | 6 (6) | 1 (1) | 1 (1) | 1 (1)
Mucosal inflammation (General disorders) | 2 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 16 (25) | 15 (27) | 6 (6) | 4 (6) | 4 (4)
Headache (Nervous system disorders) | 6 (7) | 6 (6) | 3 (5) | 2 (3) | 1 (1)
Dizziness (Nervous system disorders) | 4 (6) | 8 (9) | 1 (1) | 2 (2) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 4 (11) | 8 (14) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 4 (6) | 5 (5) | 2 (2) | 1 (1) | 2 (2)
Restless legs syndrome (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 9 (12) | 0 (0) | 3 (3) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (7) | 1 (1) | 1 (1) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 7 (10) | 10 (15) | 2 (2) | 2 (2) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 9 (11) | 2 (3) | 2 (3) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (10) | 5 (8) | 1 (1) | 2 (3) | 2 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (8) | 0 (0) | 1 (2) | 1 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 2 (6) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Ear and labyrinth disorders) | 1 (1) | 3 (11) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 10 (27) | 7 (20) | 4 (5) | 4 (4) | 2 (4)
Anaemia (Blood and lymphatic system disorders) | 9 (26) | 7 (20) | 2 (5) | 3 (8) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (20) | 3 (19) | 2 (2) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (13) | 4 (16) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 4 (4) | 1 (1) | 1 (1) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (7) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 5 (8) | 5 (7) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Oral candidiasis (Infections and infestations) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 7 (7) | 8 (8) | 2 (2) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 4 (5) | 0 (0) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 10 (16) | 8 (13) | 1 (1) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (3) | 0 (0) | 1 (2) | 1 (2) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 6 (9) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 8 (9) | 4 (4) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Vascular disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 3 (5) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 4 (5) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 3 (4) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2015-08-10): https://cdn.clinicaltrials.gov/large-docs/12/NCT01925612/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-19): https://cdn.clinicaltrials.gov/large-docs/12/NCT01925612/SAP_001.pdf